CLINICAL TRIAL: NCT04490499
Title: A Hepatitis B Vaccine Challenge Study to Demonstrate the Durability of Protection Against Hepatitis B Virus Infection in Healthy Children Vaccinated Approximately 9 Years Previously With a 2- or 3-Dose Infant Series and Toddler Dose of Vaxelis®
Brief Title: A Hepatitis B Vaccine Challenge Study After Previous Vaxelis® Vaccination (V419-013)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V419-013; V419-013 (Other: Merck); 2020-000126-26 (EudraCT Number)
Record Dates: First submitted 2020-07-28; First posted 2020-07-29 (Actual); Results first posted 2021-09-05 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Hepatitis B Vaccines; Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- HBVAXPRO™ (Experimental): Healthy children vaccinated approximately 8-9 years previously with a 2- or 3-dose infant series and toddler dose of Vaxelis® who will receive a single dose of Hepatitis B vaccine challenge (HBVAXPRO™).
  Interventions: Biological: HBVAXPRO™

INTERVENTIONS:
Biological: HBVAXPRO™ — Single 0.5 mL intramuscular dose
  Other Names: Hepatitis B virus (HBV) vaccine; V232

SUMMARY:
The purpose of this study is to demonstrate the durability of protection against hepatitis B virus (HBV) infection approximately 8-9 years after vaccination with Vaxelis®. This is an estimation study, and no formal hypothesis testing was performed.

ELIGIBILITY:
Inclusion Criteria:

* Is healthy (based on a review of medical history and targeted physical examination) based on the clinical judgment of the investigator.
* Has participated in Protocol V419-007 and received a 3 + 1 Vaxelis® schedule or participated in Protocol V419-008 and received a 2 + 1 Vaxelis® schedule.
* The participant (or legally acceptable representative if applicable) provides written informed consent/assent for the study.

Exclusion Criteria:

* Has a history of diagnosis (clinical, serological, or microbiological) of HBV infection.
* Has a known or suspected impairment of immunological function (e.g., human immunodeficiency virus (HIV), splenectomy).
* Has a known hypersensitivity to any component of the study vaccine.
* Has a known or suspected blood dyscrasias, leukemia, lymphomas of any type or other malignant neoplasms affecting the haematopoietic and lymphatic system.
* Has a bleeding disorder contraindicating intramuscular vaccinations.
* Has received any hepatitis B vaccine after participation in Protocol V419-007 or V419-008.
* Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling, or child) who is investigational site or Sponsor staff directly involved with this study.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 207 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2020-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (10):
- Finland (10):
  - Tampereen yliopisto Kokkolan rokotetutkimusklinikka ( Site 0009), Kokkola, Keski-Pohjanmaa
  - Tampereen yliopisto Oulun rokotetutkimusklinikka ( Site 0004), Oulu, North Ostrobothnia
  - Tampereen yliopisto - Tampereen rokotetutkimusklinikka ( Site 0001), Tampere, Pirkanmaa
  - Seinajoki Vaccine Research Center ( Site 0010), Seinajoki, Pohjanmaa
  - Porin rokotetutkimusklinikka ( Site 0008), Pori, Satakunta
  - Tampereen yliopisto Turun rokotetutkimusklinikka ( Site 0002), Turku, Southwest Finland
  - Tampereen yliopisto Espoon rokotetutkimusklinikka ( Site 0007), Espoo, Uusimaa
  - Tampereen yliopisto Etelä-Helsingin rokotetutkimusklinikka ( Site 0005), Helsinki, Uusimaa
  - Ita-Helsingin Rokotetutkimuskeskus ( Site 0006), Helsinki, Uusimaa
  - Tampereen yliopisto Järvenpään rokotetutkimusklinikka ( Site 0003), Jarvenpaa, Uusimaa

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Ahonen A, Zhang Y, Marcek T, Lumley J, Johnson DR, Guris D, Wilck MB. Demonstration of durable hepatitis B immune memory in children vaccinated with a DTaP5-IPV-HepB-Hib infant-toddler series 7 to 8 years previously. Hum Vaccin Immunother. 2022 Nov 30;18(5):2073747. doi: 10.1080/21645515.2022.2073747. Epub 2022 Jun 2. PMID 35653552

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Approximately 200 planned to be enrolled and 207 were enrolled.
Groups:
- HBVAXPRO™: Healthy children vaccinated approximately 8-9 years previously with a 2- or 3-dose infant series and toddler dose of Vaxelis® who received a single dose of Hepatitis B vaccine challenge (HBVAXPRO™).
Period: Overall Study
Arm/Group | HBVAXPRO™
Started | 207
Vaccinated | 205
Completed | 205
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | HBVAXPRO™
Number analyzed (Participants) | 207
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.4 (0.5) [lower limit 0.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97
  Male | 110
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 205
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 205
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Finland | 207

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Protective Hepatitis B Surface Antibody Level of ≥10 Milli International Units/mL (mIU/mL) at 30 Days Post-Challenge With HBVAXPRO™
Description: Participant serum samples were collected for analysis with an enhanced chemiluminescence (ECi) assay to determine the concentration of antibodies to hepatitis B surface antigen (HBsAg). Response rate was the percentage of participants with a protective hepatitis B surface antibody (anti-HBs) level of ≥ 10 mIU/mL at Day 30 post-challenge.
Time Frame: Day 30
Population: The analysis population consisted of all enrolled participants without deviations from the protocol (i.e., did not receive study vaccine, use of prohibited medicine/vaccine, or blood sample collected outside of analysis window) that may substantially affect the results of the immunogenicity endpoint.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | HBVAXPRO™
Number analyzed (Participants) | 202
Percentage of Participants | 99.5 (97.3) [97.3 to 100.0]

2. Secondary Outcome: Geometric Mean Concentration of Antibodies to Hepatitis B Surface Antigen
Description: Participant serum samples will be assessed with an ECi assay for anti-HBs geometric mean concentrations (GMCs) pre-challenge on Day 1 and 30 days post-challenge with HBVAXPRO™ in mIU/mL.
Time Frame: Day 1 and Day 30
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | HBVAXPRO™
Number analyzed (Participants) | 205
mIU/mL
  Day 1 Pre-challenge | 9.63 [7.88 to 11.76]
  Day 30 Post-challenge: number analyzed (Participants) | 202
  Day 30 Post-challenge | 685.84 [605.67 to 776.63]

ADVERSE EVENTS:
Time Frame: Up to Day 30
Description: The analysis population included all participants who received study vaccine and had safety follow-up data after the vaccination. The all-cause mortality analysis population included all enrolled participants. Per protocol, reported non-serious adverse events only include non-serious adverse events that lead to study discontinuation.
Arm/Group | HBVAXPRO™
All-Cause Mortality (participants affected / at risk) | 0/207
Serious Adverse Events (participants affected / at risk) | 0/205
Other Adverse Events (participants affected / at risk) | 0/205

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/99/NCT04490499/Prot_SAP_000.pdf